CLINICAL TRIAL: NCT04457960
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single and Multiple Ascending Dose Study in Healthy Participants and Multiple Dose Study in Participants With Ulcerative Colitis to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of JNJ-66525433
Brief Title: A Study of JNJ-66525433 in Healthy Participants and Participants With Ulcerative Colitis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Decision.
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: CR108764; 2018-003743-29 (EudraCT Number); 66525433IBD1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2020-07-01; First posted 2020-07-07 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy; Colitis, Ulcerative
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- JNJ-66525433 (Experimental): Participants will receive JNJ-66525433 in increasing dose level 1 to dose level 4 in Parts 1, 2, and dose level 3 in part 3.
  Interventions: Drug: JNJ-66525433
- Placebo (Placebo Comparator): Participants will receive matching placebo in Parts 1, 2 and 3.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JNJ-66525433 — Participants will receive JNJ-66525433 oral capsules.
  Arms: JNJ-66525433
Drug: Placebo — Participants will receive matching placebo oral capsules.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate safety and tolerability of JNJ 66525433 compared with placebo after administration of: 1) single ascending oral doses of JNJ 66525433 administered to healthy participants (Part 1), 2) multiple, ascending oral doses of JNJ 66525433, administered to healthy participants once daily over 14 consecutive days (Part 2), and 3) multiple oral doses of JNJ 66525433, administered once daily over 14 consecutive and once daily over 42 consecutive days in participants with ulcerative colitis (UC) (Part 3).

ELIGIBILITY:
Inclusion Criteria:

For Part 1 and Part 2, healthy volunteers

* Have a body mass index (BMI) between 18 and 30 kilogram per meter square (kg/m^2) (BMI = weight/height), inclusive, and a body weight of no less than 50 kilogram (kg) and maximum weight of 100 kg
* Have normal bowel movements, ranging from 1 to 3 times daily to every other day and have normal consistencies according to the Bristol Stool Scale, ranging from 3 to 5 at admission

For Part 3, participants with ulcerative colitis (UC)

* Have a clinical diagnosis of UC at least 3 months before screening
* Have moderately to severely active UC, defined as a Week 0 mayo score of 6 to 12, inclusive, based on central read of the video endoscopy performed during the screening
* Have a greater than or equal to (>=) 2 endoscopy subscore of the Week 0 mayo score based on central read of the video endoscopy performed during the screening

Exclusion Criteria:

For Part 1 and Part 2, healthy volunteers

* History of liver or renal insufficiency, significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances
* Known allergies, hypersensitivity, or intolerance to antisense oligonucleotides, JNJ-66525433 or its excipients

For Part 3, participants with UC

* Has UC limited to the rectum only or to <20 centimeter (cm) of the colon evaluated by endoscopy at screening
* Presence of a stoma
* Presence or history of a fistula at any time

COVID-related

* If a participant is excluded due to recent Coronavirus disease (COVID-19) related features, the reason for screen failure should be documented in the case report form under the exclusion criterion of having a condition for which participation would not be in the participant's interest or could confound study assessments
* The field of COVID-related testing (for presence of, and immunity to, the severe acute respiratory syndrome coronavirus 2 [SARS-CoV-2] virus) is rapidly evolving. Additional testing may be performed as part of screening and/or during the study if deemed necessary by the investigator and in accordance with current regulations / guidance from authorities / standards of care

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-10-13 (Actual); Study Completion 2021-10-13 (Actual)

PRIMARY OUTCOMES:
Part 1, 2 and 3: Number of Participants with Treatment-emergent Adverse Events (TEAEs) as a Measure of Safety and Tolerability | Up to 224 Days
  An adverse event (AE) is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. Any AE occurring at or after the initial administration of study intervention through the day of last dose plus 30 days will be considered as TEAE.
Part 1, 2 and 3: Number of Participants with Vital Sign Abnormalities | Up to 224 Days
  Number of participants with vital sign abnormalities (temperature), pulse/heart rate, respiratory rate and blood pressure) will be reported.
Part 1, 2 and 3: Number of Participants with Physical Examination Abnormalities | Up to 224 Days
  Number of participants with physical examination abnormalities will be reported.
Part 1, 2 and 3: Number of Participants with Hematology Laboratory Abnormalities | Up to 224 Days
  Number of participants with hematology laboratory abnormalities will be reported.
Part 1, 2 and 3: Number of Participants with Chemistry Laboratory Abnormalities | Up to 224 Days
  Number of participants with chemistry laboratory abnormalities will be reported.
Part 1, 2 and 3: Number of Participants with Urinalysis Laboratory Abnormalities | Up to 224 Days
  Number of participants with abnormalities in urinalysis will be reported.
Part 2 and 3: Number of Participants with Abnormalities in High Sensitivity C- Reactive Protein (hs-CRP) | Up to 224 Days
  Number of participants with abnormalities in hs-CRP will be reported using a validated, high sensitivity CRP assay.
Part 2 and 3: Number of Participants with Abnormalities in Fecal Calprotectin | Up to 224 Days
  Assays for fecal calprotectin will be performed using a validated method.
Part 2 and 3: Incidence of Enteric Pathogens in Stool Samples | Up to 224 Days
  Stool culture and Clostridium difficile toxin assay will be used for enteric pathogen assessment.
Part 1, 2 and 3: Number of Participants with Electrocardiogram (ECG) Abnormalities | Up to 224 Days
  Number of participants with ECG abnormalities will be reported.

SECONDARY OUTCOMES:
Part 1, 2 and 3: Plasma Concentrations of JNJ-66525433 | Up to 224 Days
  Plasma concentrations of JNJ-66525433 will be reported.
Part 1: Plasma Concentrations of JNJ-66525433 After Fasted or Fed Dosing | Up to Day 14
  Plasma concentrations of JNJ-66525433 after fasted or fed dosing will be reported.
Part 3: Mayo Score | Up to Day 84
  Mayo scoring system is used for assessment of ulcerative colitis activity. The Mayo score consists of 4 subscores (stool frequency, rectal bleeding, physician's global assessment, and endoscopy findings) each ranges from 0 to 3. The Mayo score is calculated as the sum of these 4 subscores and can range between 0 and 12, where higher score indicates severe disease.
Part 3: Partial Mayo Score | Up to Day 70
  Partial Mayo score is calculated as the sum of 3 subscores (stool frequency, rectal bleeding, and physician's global assessment) and ranges from 0 to 9 points. Higher score indicates severe disease.
Part 3: Endoscopic Subscore | Up to Day 84
  Endoscopy sub-score ranges from 0 to 3 where; 0 = normal or inactive disease; 1 = mild disease (erythema, decreased vascular pattern, mild friability); 2 = moderate disease (marked erythema, absent vascular pattern, friability, erosions); 3 = severe disease (spontaneous bleeding, ulceration).
Part 3: Inflammatory Bowel Disease Questionnaire (IBDQ) Total Score | Days 1, 7, 14, 28, 43, 70 and 84
  IBDQ18 is a validated, 32-item, self-reported questionnaire for participants with inflammatory bowel disease (IBD) that will be used to evaluate the disease-specific health-related quality of life across 4 dimensional scores: bowel symptoms (loose stools, abdominal pain), systemic functions (fatigue, altered sleep pattern), social function (work attendance, need to cancel social events), and emotional function (anger, depression, irritability). Scores range from 32 to 224, with higher scores indicating better outcomes.
Part 2 and 3: Target Engagement of Messenger Ribonucleic Acid (mRNA) Levels | Up to 182 Days
  Levels of mRNA knockdown will be reported to assess target engagement in biopsy tissue by dose level over time.
Part 2 and 3: Tissue Biopsy JNJ-66525433 Concentrations | Up to 182 Days
  Tissue biopsy concentrations of JNJ-66525433 will be reported.
Plasma Concentrations of JNJ-66525433 After Two Meal Timing Conditions | Up to 22 Days
  Plasma concentrations of JNJ-66525433 after two meal timing condition (fed state to modified fasted state) will be reported (if conducted).
Faecal Concentrations of JNJ-66525433 After Two Meal Timing Conditions | Predose, up to 120 hours postdose
  Stool assessment will be done to characterize the presence of JNJ-66525433 after two meal timing conditions (fed state to modified fasted state) will be reported (if conducted).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Charite Research Organisation GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency